CLINICAL TRIAL: NCT06099743
Title: An ACT-Based Supportive Intervention for Patients With Central Nervous System Tumors
Brief Title: ASCENT Intervention for Brain Tumor Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Deborah A Forst, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-436
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Malignant Brain Tumor; Glioma; Coping Skills; Distress, Emotional
Keywords: glioma; supportive care; brain tumor; psychological distress; support
MeSH Terms: conditions — Brain Neoplasms; Glioma | interventions — Psychosocial Intervention

STUDY DESIGN:
Intervention Model Description: In this pilot randomized control trial (n=100) participants will be randomized 1:1 to the intervention versus usual care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pilot RCT: ASCENT Arm (Experimental): Enrolled patients will receive an intervention manual and will participate in six weekly or biweekly individual sessions with a clinician (e.g. nurse or behavioral health specialist).
  Participants will be asked to complete surveys at baseline, 6 weeks, 12 weeks, and 16 weeks.
  Interventions: Behavioral: Psychosocial intervention
- Pilot RCT: Control Arm (Active Comparator): Participants will receive usual supportive care, which includes referral to cancer center supportive care services (e.g., social work) upon request from the patient, caregiver, or clinician.
  Participants will be asked to complete surveys at baseline, 6 weeks, 12 weeks, and 16 weeks.
  Interventions: Other: Usual supportive care

INTERVENTIONS:
Behavioral: Psychosocial intervention — Intervention manual and six one-on-one coaching sessions.
  Other Names: ASCENT
  Arms: Pilot RCT: ASCENT Arm
Other: Usual supportive care — Referral to cancer center supportive care services (e.g., social work) as needed, upon request from the patient, caregiver, or clinician.
  Arms: Pilot RCT: Control Arm

SUMMARY:
The goal of this study is to refine and test a psychosocial intervention called ASCENT (ACT-based Supportive intervention for patients with CENTral nervous system tumors). This intervention was developed to help patients after being diagnosed with a brain tumor. The main question this study aims to answer is whether this intervention is feasible (i.e., possible to carry out) and acceptable (i.e., considered helpful) to patients. Participants will be asked to take part in 6 coaching sessions and complete short surveys at four different time points. Some participants will be asked to share feedback via interviews.

DETAILED DESCRIPTION:
This study will examine the feasibility and acceptability of a novel, population-specific intervention designed to help patients with newly diagnosed malignant brain tumors cope with their illness.

This project is currently recruiting participants for intervention refinement activities in preparation for the pilot RCT. For intervention refinement, we are enrolling 15 stakeholders and 10 open pilot participants to gather feedback about the intervention to improve it prior to commencing the randomized controlled trial. The stakeholder feedback and open pilot refinement phase of the study is critical for intervention refinement for the RCT. The investigators will then evaluate the feasibility and acceptability of the refined ASCENT intervention versus usual care in this pilot randomized controlled trial (n=100). The investigators will also estimate preliminary effects of ASCENT on psychological and behavioral outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Massachusetts General Hospital Cancer Center Patient
* Within 6 months of diagnosis of malignant primary Central Nervous System (CNS) tumor
* English speaking

Exclusion Criteria:

* Inability to provide informed consent as assessed by the study team (e.g., due to severe cognitive impairment/dementia)
* Moderate to severe receptive aphasia (Quick Aphasia Battery sentence comprehension subscale < 8)
* Current or imminent hospice enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Intervention: Percentage of Eligible Patients Who Enroll and Participate in the Intervention | Up to 12 weeks
  The investigators will assess feasibility by examining the percentage of eligible patients who agree to enroll in the study and the percentage of enrolled patients who participate in all six intervention sessions. The intervention will be deemed feasible if at least 60% of eligible patients enroll in the study and if at least 70% of enrolled patients complete at least half of the sessions.
Acceptability of the Intervention: Percentage of Participants who Have High Satisfaction with the Intervention | 12 weeks
  The investigators will assess acceptability via examining the distribution of patient scores for the 8-item Client Satisfaction Questionnaire (CSQ-8). CSQ-8 scores range from 8 to 32, with higher scores indicating higher satisfaction. The intervention will be deemed acceptable if at least 70% of patients score at least 24 points on the CSQ-8.

SECONDARY OUTCOMES:
Exploratory: Coping Skills | Up to 16 weeks
  The investigators will explore the effect of ASCENT on coping skills using the Measure of Current Status (MOCS) Part A. The MOCS Part A is a 13-item measure of self-perceived coping skills with scores ranging from 0-52 with higher scores indicating higher self-perceived coping skills.
Exploratory: Values-driven behavior | Up to 16 weeks
  The investigators will explore the effect of the ASCENT intervention on values driven behavior using the Valued Living Questionnaire (VLQ). In this questionnaire, respondents rate the importance of 10 domains of living and their consistency living in accordance with those values in the past week. Scores range from 10-100 with higher scores indicating a value with more importance.
Exploratory: Prognostic distress | Up to 16 weeks
  The investigators will explore the effect of the ASCENT intervention on prognostic awareness using the Prognostic Awareness Impact Scale (PAIS). This 34-item questionnaire measures three domains: cognitive understanding of prognosis, emotional coping with prognosis, and adaptive response (i.e., the capacity to use prognostic awareness to inform life decisions). The cognitive understanding domain consists of two items including a question asking patients if their oncologist has said that their cancer is curable and a question asking patients to report the likelihood that they would be cured of their cancer, assessed on a 7-point scale ranging from no chance/0% to extremely likely/>90%. The emotional coping domain consists of eight items, with a score range of 0-24, with higher scores indicating better emotional coping with prognosis. The adaptive response domain consists of 12 items, with a score range of 0-36, with higher scores indicating better adaptive response to prognosis
Exploratory: Depression symptoms | Up to 16 weeks
  The investigators will explore the effect of the ASCENT intervention on depression symptoms using the Patient Health Questionnaire -8 (PHQ-8) The PHQ-8 is an 8 item measure with scores ranging from 0-24 and higher scores indicating more severe depression.
Exploratory: Quality of Life | Up to 16 weeks
  The investigators will explore the effect of ASCENT on symptom burden and quality of life using the Functional Assessment of Cancer Therapy - Brain (FACT-Br). The FACT-Br is a 50-item tool consisting of four subscales assessing well-being across four domains (physical, functional, emotional, and social), as well as additional questions specific to patients with brain tumors. Scores range from 0-200 with higher scores indicating better health-related quality of life.
Exploratory: Loneliness | Up to 16 weeks
  The investigators will explore the effect of ASCENT on loneliness and social isolation using the 20 item UCLA Loneliness Scale with scores ranging from 20-80 and higher scores indicating more loneliness.
Exploratory: Anxiety symptoms | Up to 16 weeks
  The investigators will explore the effect of the ASCENT intervention on depression symptoms using the Generalized Anxiety Disorder - 7 (GAD-7) questionnaire. The GAD-7 has scores ranging from 0-21 with higher scores indicating more severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Forst, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available to the public via openICPSR (Inter-University Consortium for Political and Social Research).
  Raw interview data may contain potentially identifiable contextual material, the study will not share raw interview data to preserve confidentiality. All other data (de-identified demographic information, de-identified clinical data, participant survey responses, and coded interview data) will be preserved and shared. Respondent identifiers will not be shared.
  Data to be made publicly available will include the study protocol, the semi-structured exit interview guide, data collection instruments, and a codebook describing relevant features of measured variables (e.g., variable name, related survey questions and possible responses, codes for missing values). The codebook will be accompanied by univariate descriptive statistics for variables. A User Guide will be made accessible with descriptions of data and instructions for interpretation.
Supporting Information: Study Protocol
Time Frame: In accordance with the National Cancer Institute's Clinical Trial Access Policy, results will be made publicly accessible within 12 months of the study completion date or 12 months of final subject data collection (whichever comes first).
  Data will remain available for as long as the repository is in existence.
Access Criteria: Deidentified participant data will be made available to the public via openICPSR (Inter-University Consortium for Political and Social Research). However, any member of the public wishing to gain access to this data must create an account with ICPSR and therefore agree to its Terms of Use designed to protect study participants and limit redistribution of the downloaded dataset.